CLINICAL TRIAL: NCT03198091
Title: An Open Label, Single Arm, Multiple Center Study Observing the Efficacy of Dun Ye Guan Xin Ning Tablet in Patients With Coronary Artery Disease of Angina Pectoris
Brief Title: Efficacy of Dun Ye Guan Xin Ning Tablet in Patients With Stable Angina Pectoris
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Collaborators: Jiangsu Wanbang Pharmaceutical Marketing Co.,Ltd. (Unknown)
Responsible Party: Principal Investigator, Yong Huo, Director of the Department of Cardiology and heart center of Peking University First Hospital, Peking University First Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DY-SH-1601
Record Dates: First submitted 2017-05-25; First posted 2017-06-23 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Coronary Heart Disease
Keywords: stable angina pectoris; Dun Ye Guan Xin Ning
MeSH Terms: conditions — Coronary Disease; Angina, Stable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dun Ye Guan Xin Ning mono-therapy (Experimental)
  Interventions: Drug: Dun Ye Guan Xin Ning

INTERVENTIONS:
Drug: Dun Ye Guan Xin Ning — Dun Ye Guan Xin Ning tablet 320 mg orally every time and 3 times per day for 6 months.

SUMMARY:
This registry is designed to investigate factors affecting the efficacy of Dun Ye Guan Xin Ning tablet on patients with stable angina. The potential hypothesis is that Dun Ye Guan Xin Ning has a better effect on different subgroup patients with certain characteristics.

DETAILED DESCRIPTION:
A total of 1000 eligible patients enrolled from 20 centers will take standard medications of care for stable angina plus Dun Ye Guan Xin Ning tablet for 6 months. Symptoms, questionnaires (SAQ, PSQI, and angina pectoris quantitative table of Chinese medicine symptoms scale), lipid, fasting glucose, homocysteine, EKG, blood pressure and other physical examination will be collected at baseline and follow-up. Among them, 200 patients will measure and inflammation biomarkers and endothelial function for further evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 75 years.
2. Documented stable angina pectoris.
3. During a period of time (more than 3 months), the duration, severity and the threshold of angina is relatively stable.
4. Patients with at least one of the following events: ① patients who have done PCI or CABG for more than half a year; ② coronary CTA angiography or coronary angiography showed at least one major coronary artery stenosis ≥ 50%. Symptom occurs at least once per month.
5. Medications remain stable within 1 month before the enrollment.
6. Patients have the ability to understand the study, and can cooperate with researchers to carry out the test.
7. Signed inform consent.

Exclusion Criteria:

1. Patents with coronary heart disease acute coronary syndrome during the last 6 months.
2. Patients with aortic stenosis, hypertrophic cardiomyopathy and other diseases leading to angina.
3. Patients have other heart disease, severe neurosis, menopausal syndrome, hyperthyroidism, cervical spondylosis, biliary heart disease, gastroesophageal reflux caused by chest pain.
4. Patients combined with severe cardiopulmonary insufficiency (NYHA grade III ord IV), pulmonary insufficiency graded reference COPD clinical severity of lung function grade III (FEV1 / FVC <70%, 30% 1 / FVC% of predicted value <50%) and grade IV), severe arrhythmia (eg. III degree atrioventricular block)
5. Patients combined with liver, kidney, hematopoietic system and other serious primary disease patients (TBil ≥ 1.5ULN, AST ≥ 2ULN, ALT ≥ 2ULN, serum creatinine ≥ 1.5ULN, Hb <9mg/dL).
6. Patients with cognitive, intellectual, or mental disorders.
7. Those who can not take oral medication.
8. Allergy to any component of this product.
9. Patients received the trial medication within 28 days prior to the first treatment of this product.
10. Lactating or pregnant women.
11. Patients who are unwilling or unable to contraceptive in the reproductive period.
12. Poor medication compliance.
13. Other circumstances that the investigator considers unsuitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2017-03-30 (Actual); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Angina pectoris symptom | 6 month
  Improvement od angina pectoris symptom

SECONDARY OUTCOMES:
Life quality | 6 month
  using seattle Angina Questionnaire
Sleep quality | 6 month
  using pittsburgh sleep quality index
Chest tightness | 0, 1 month, 3 month, 6 month
  using angina pectoris quantitative table of Chinese medicine symptoms
Biomarkers | 6 month
  levels of TG，TC, LDL, HDL, HCY, IL-6、TNF-α、and CRP

OTHER OUTCOMES:
Vascular endothelial function | 0, 1 month, 3 month, 6 month
  using ZX7M-Endo-pat2000

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No